CLINICAL TRIAL: NCT05289180
Title: A Novel Method for Cardiac Allograft Monitoring:Transbrachial Right Ventricle Endomyocardial Biopsy
Brief Title: Brachial Right Ventricle - Endomyocardial Biopsy
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-01132
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants undergoing Heart Catherization: Participants undergoing Heart Catherization and will complete a research survey focusing on the comfort and anxiety during procedure. Participants will be followed for 18 months after enrollment. For each clinically indicated Brachial RV-EMB Biopsy during the 18-month follow up period, data from biopsy and pre and post-procedure echocardiograms will be reviewed and recorded for research purposes. A post-procedure questionnaire and post-discharge phone call will also take place after each procedure.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — A questionnaire will be administered post-procedure to assess for pain and anxiety. This questionnaire will be administered by study personnel delegated to administer questionnaires, namely the study coordinator or PI.

SUMMARY:
This is an observational study that will recruit NYU Langone patients undergoing standard of care right ventricle endomyocardial biopsy. Patients who undergo planned RV-EMB via transbrachial access will be invited to take part in the study.

DETAILED DESCRIPTION:
Data including severity of tricuspid regurgitation and tamponade from pre and post procedure bedside echocardiograms, total procedure duration, radiation exposure and fluoroscopy time, sedatives used (if any) and bleeding/hematoma formation (if any) will be collected. A post-procedural survey will be administered to patients by study staff to assess comfort level and anxiety during procedure. A post procedure phone call will take place 3-5 days after procedure to assess for bruising, swelling or bleeding at the site of Brachial RV-EMB.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 90 years old
* Patient is undergoing standard of care right heart catheterization with endomyocardial biopsy
* Patient has right arm brachial access available
* Patient is willing and able to provide written informed consent.

Exclusion Criteria:

* Peripherally inserted central catheter (PICC) line or arteriovenous (AV) fistula
* Severe untreated tricuspid valve regurgitation
* Female patients who are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Right heart endomyocardial biopsy is classically approached via jugular or femoral access. Brachial access has not been widely studied and appears to be an efficient and safe method for performing endomyocardial biopsies. We hypothesize that transbrachial right endomyocardial biopsy is a safe, comfortable and equally effective procedure to endomyocardial biopsies via classical access methods. This single arm study will focus on brachial endomyocardial biopsy and will be compared with historical data.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction in Right endomyocardial biopsy via brachial access | Day 1 to Day 540
  Assessed by patients self report of their experience when undergoing right endomyocardial biopsy via brachial access compared to transjugular and transfemoral right ventricle endomyocardial biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Tajinderpal Saraon, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Tajinderpal.Saraon@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.